CLINICAL TRIAL: NCT05046379
Title: Lipidomics for Identification of New Biomarkers for Fabry Disease
Brief Title: Studying Lipids as Potential Biomarkers in Patients With Fabry Disease
Status: Completed | Type: Observational
Sponsor: Vastra Gotaland Region (Other Government)
Collaborators: Karolinska University Hospital (Other); Uppsala University Hospital (Other); Sahlgrenska University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: Lipidomics in Fabry
Record Dates: First submitted 2021-09-06; First posted 2021-09-16 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-04

CONDITIONS: Fabry Disease
Keywords: Biomarkers; Fabry disease; Lipidomics
MeSH Terms: conditions — Fabry Disease

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Biobank Väst
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with Fabry disease: Adult men and women with well characterized Fabry disease
  Interventions: Other: Lipidomics
- Healthy controls (with no Fabry disease): Adult men and women from the endocrinology and nephrology in- or out-patient clinic
  Interventions: Other: Lipidomics

INTERVENTIONS:
Other: Lipidomics — Lipidomics is the large-scale study of lipids (fats and fat-like molecules) within biological systems. It involves identifying and quantifying the wide variety of lipids in cells, tissues, or organisms to understand their roles in metabolism, signaling, and disease. Lipidomics is a subfield of metabolomics and uses advanced analytical techniques, like mass spectrometry, to profile lipid molecules. It helps in studying how lipids contribute to cellular functions, disease development, and responses to therapies.

SUMMARY:
Compare levels of lipids between well characterised enzymatically-genetically-phenotypically patients with Fabry disease and healthy controls (with no Fabry disease).

Correlate levels of lipids in patients with Fabry disease to clinical outcomes/manifestations of the disease.

DETAILED DESCRIPTION:
The hypothesis is that Sphingosine-1 Phosphate (S1P) or any other related sphingoid bases and/or other lipid class could be a marker of the severity of cardiovascular remodelling in Fabry disease.

The overall approach is, by minimising possible pre-analytical and analytical biases, to study by lipidomics in well characterised enzymatically, genetically and phenotypically patients with Fabry disease, if S1P or any other lipid (including other glycosphingolipids) is shown to be a biomarker for the diagnosis, monitoring of disease activity and prognosis (including cardiovascular outcomes).

ELIGIBILITY:
Inclusion criteria for cases:

* Adult men and women
* Well characterized Fabry disease in terms of i. alpha-Gal A enzyme activity, ii. mutation in alpha-Gal A (GLA) gene, and iii. disease manifestations
* Followed at one of the 3 centers for patients with Fabry disease in Sweden (Karolinska in Stockholm, Sahlgrenska in Gothenburg, Akademiska in Uppsala)

Signed informed consent prior to sample collection is mandatory for inclusion to the study.

Inclusion criteria for controls:

* Adult men and women
* Followed/treated at the endocrinology or nephrology in- or out-patient clinic at Sahlgrenska University Hospital in Gothenburg
* Matched for age, sex, estimated Glomerular filtration rate (eGFR) with the cases with Fabry disease

Exclusion criteria for controls:

* Fabry disease
* Liver disease with elevated transaminases
* Ongoing infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult men and women with well characterized Fabry disease and adult men and women with no Fabry disease and liver disease with elevated transaminases and ongoing infection.
Sampling Method: Non-Probability Sample
Enrollment: 108 (Actual)
Dates: Start 2021-10-14 (Actual); Primary Completion 2024-04-28 (Actual); Study Completion 2024-04-28 (Actual)

PRIMARY OUTCOMES:
Lipidomics | Samples are going be collected during 1 year at the fasting state in the morning. At a random day in both Fabry patients with no treatment and cases. Up to 24 hours before next treatment in Fabry patients with ongoing treatment.
  Lipid species from several lipid classes

CONTACTS AND LOCATIONS:
Overall Officials: Maria Blomqvist, Ass.Prof., Principal Investigator — Västra Götalandsregion
Locations (3):
- Sweden (3):
  - Sahlgrenska University Hospital, Gothenburg
  - Karolinska University Hospital, Stockholm
  - Akademiska University Hospital, Uppsala

IPD SHARING:
Plan to Share IPD: No